CLINICAL TRIAL: NCT06427954
Title: Randomized Trial of Mobile Application to Improve Health-Related Outcomes in Patients With Advanced Lung Cancer
Brief Title: Mobile Application to Improve Health-Related Outcomes in Patients With Advanced Lung Cancer
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-091
Record Dates: First submitted 2024-05-17; First posted 2024-05-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
Keywords: Quality of life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE Digital Health App (Active Comparator): Patients assigned to the intervention will be provided a study-issued tablet computer from which they will access the THRIVE digital health app. Study staff will give intervention patients a comprehensive tutorial and detailed instructions regarding how to use the app. Tutorial sessions may be conducted in person during a clinic appointment, via telephone, and/or via Zoom videoconferencing. Participants will complete the intervention modules at their desired pace over approximately 10 weeks.
  Interventions: Behavioral: Digital Health App
- Usual Care (No Intervention): Patients assigned to the usual care group will not receive the digital app but rather standard oncology care.

INTERVENTIONS:
Behavioral: Digital Health App — access to a digital health app
  Arms: THRIVE Digital Health App

SUMMARY:
Multi-site randomized trial of the THRIVE digital health application versus usual care to evaluate the effect of THRIVE on quality of life (QOL), physical and psychological symptoms, coping, and self-efficacy in 250 patients with newly diagnosed advanced lung cancer.

DETAILED DESCRIPTION:
Multi-site randomized controlled trial of the THRIVE digital health application versus usual care in 250 patients diagnosed with advanced lung cancer within the previous 12 weeks to examine the effect of the intervention on patient-reported QOL, physical symptoms, anxiety and depression symptoms, coping, and self-efficacy. Participants will be randomized in a 1:1 fashion and stratified by study site and lung cancer type to ensure a balanced representation of these factors between the two study groups. The study team will provide iPads to patients assigned to THRIVE and provide instructions on how to use the iPad and digital app. The study team will administer patient-reported outcome measures at enrollment and again at six, 12, and 24 weeks post-enrollment to evaluate the short and long-term impact of THRIVE.

ELIGIBILITY:
Inclusion Criteria:

* Adults (greater than or equal to 18 years)
* Diagnosed with advanced non-small cell lung cancer (NSCLC) that is not being treated with curative intent or extensive stage small cell lung cancer (SCLC) within the past 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) = 0-2 (i.e., fully active to at least ambulatory and up and about more than 50% of waking hours).
* Sufficient English proficiency to utilize THRIVE in English (Note: patients can complete outcome measures in Spanish if preferred).

Exclusion Criteria:

* Significant uncontrolled psychiatric disorder (e.g., psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (e.g., dementia, cognitive impairment), which the treating oncology clinician reports would prohibit the ability to participate in study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Lung (FACT-L) | 12 weeks
  Quality of Life (higher scores indicate better quality of life)

SECONDARY OUTCOMES:
MD Anderson Symptom Inventory (MDASI) | 12 weeks
  Physical Symptoms (higher scores indicate worse symptoms)
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Anxiety and Depression Symptoms (higher scores indicate worse symptoms)

OTHER OUTCOMES:
Brief Cope (Modified) | 12 weeks
  Coping (higher scores indicate greater use of coping strategy)
Cancer Self-Efficacy Scale | 12 weeks
  Self-efficacy (higher scores indicate greater self-efficacy)
FACT-L | Over 24 weeks
  Quality of Life (higher scores indicate better quality of life)
MDASI | Over 24 weeks
  Physical Symptoms (higher scores indicate worse symptoms)
HADS | Over 24 weeks
  Anxiety and Depression Symptoms (higher scores indicate worse symptoms)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - Veteran Affairs Greater Los Angeles Health Care, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts